CLINICAL TRIAL: NCT05973487
Title: A Phase 1 Basket Study Evaluating the Safety and Feasibility of T-Plex, Autologous Customized T Cell Receptor-Engineered T Cells Targeting Multiple Peptide/HLA Antigens in Participants With Antigen-positive Locally Advanced (Unresectable) or Metastatic Solid Tumors
Brief Title: A Basket Study of Customized Autologous TCR-T Cell Therapies in Patients With Locally Advanced (Unresectable) or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TScan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSCAN-002
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer; Cervical Cancer; Non-small Cell Carcinoma; Melanoma; Ovarian Cancer; Anogenital Cancers; HPV - Anogenital Human Papilloma Virus Infection; HPV-Related Cervical Carcinoma; HPV-Related Carcinoma; HPV-Related Squamous Cell Carcinoma; HPV-Related Malignancy; HPV-Related Adenocarcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma; HPV-Related Adenosquamous Carcinoma; HPV-Associated Vaginal Adenocarcinoma; HPV-Related Endocervical Adenocarcinoma; HPV-Related Anal Squamous Cell Carcinoma; HPV-Related Verrucous Carcinoma; HPV-Related Penile Squamous Cell Carcinoma; HPV-Related Vulvar Squamous Cell Carcinoma; HPV Positive Rectal Squamous Cell Carcinoma
Keywords: HPV16 E7; MAGE-A1; TCR-T Therapy; Cell Therapy; Immunotherapy; TScan Therapeutics; TSCAN-002; TSCAN-003; PRAME; MAGE-C2; MAGE-A4
MeSH Terms: conditions — Head and Neck Neoplasms; Uterine Cervical Neoplasms; Melanoma; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (28):
- Monotherapy Cohort A (Experimental): TSC-204-A0201
  Interventions: Biological: TSC-204-A0201
- Monotherapy Cohort B (Experimental): TSC-204-C0702
  Interventions: Biological: TSC-204-C0702
- Monotherapy Cohort C (Experimental): TSC-200-A0201
  Interventions: Biological: TSC-200-A0201
- T-Plex Combination Cohort A + B (Experimental): TSC-204-A0201 and TSC-204-C0702
  Interventions: Biological: TSC-204-A0201 + TSC-204-C0702
- T-Plex Combination Cohort B + C (Experimental): TSC-204-C0702 and TSC-200-A0201
  Interventions: Biological: TSC-204-A0201 + TSC-200-A0201
- T-Plex Combination Cohort A + C (Experimental): TSC-204-A0201 and TSC-200-A0201
  Interventions: Biological: TSC-204-C0702 + TSC-200-A0201
- Monotherapy Cohort D (Experimental): TSC-203-A0201
  Interventions: Biological: TSC-203-A0201
- T-Plex Combination Cohort A + D (Experimental): TSC-204-A0201 + TSC-203-A0201
  Interventions: Biological: TSC-204-A0201 + TSC-203-A0201
- T-Plex Combination Cohort B + D (Experimental): TSC-204-C0702 + TSC-203-A0201
  Interventions: Biological: TSC-204-C0702 + TSC-203-A0201
- Monotherapy Cohort E (Experimental): TSC-204-A0101
  Interventions: Biological: TSC-204-A0101
- Monotherapy Cohort F (Experimental): TSC-201-B0702
  Interventions: Biological: TSC-201-B0702
- T-Plex Combination Cohort A + E (Experimental): TSC-204-A0201 + TSC-204-A0101
  Interventions: Biological: TSC-204-A0201 + TSC-204-A0101
- T-Plex Combination Cohort A + F (Experimental): TSC-204-A0201 + TSC-201-B0702
  Interventions: Biological: TSC-204-A0201 + TSC-201-B0702
- T-Plex Combination Cohort B + E (Experimental): TSC-204-C0702 + TSC-204-A0101
  Interventions: Biological: TSC-204-C0702 + TSC-204-A0101
- T-Plex Combination Cohort B + F (Experimental): TSC-204-C0702 + TSC-201B0702
  Interventions: Biological: TSC-204-C0702 + TSC-201-B0702
- T-Plex Combination Cohort C + D (Experimental): TSC-200-A0201 + TSC-203-A0201
  Interventions: Biological: TSC-200-A0201 + TSC-203-A0201
- T-Plex Combination Cohort C + E (Experimental): TSC-200-A0201 + TSC-204-A0101
  Interventions: Biological: TSC-200-A0201 + TSC-204-A0101
- T-Plex Combination Cohort C + F (Experimental): TSC-200-A0201 + TSC-201B0702
  Interventions: Biological: TSC-200-A0201 + TSC-201-B0702
- T-Plex Combination Cohort D + E (Experimental): TSC-203-A0201 + TSC-204A0101
  Interventions: Biological: TSC-203-A0201 + TSC-204-A0101
- T-Plex Combination Cohort D + F (Experimental): TSC-203-A0201 + TSC-201B0702
  Interventions: Biological: TSC-203-A0201 + TSC-201-B0702
- T-Plex Combination Cohort E + F (Experimental): TSC-204-A0101 + TSC-201-B0702
  Interventions: Biological: TSC-204-A0101; Biological: TSC-201-B0702
- Monotherapy Cohort G (Experimental): TSC-202-A0201
  Interventions: Biological: TSC-202-A0201
- T-Plex Combination Cohort A + G (Experimental): TSC-204-A0201 + TSC-202-A0201
  Interventions: Biological: TSC-204-A0201 + TSC-202-A0201
- T-Plex Combination Cohort B + G (Experimental): TSC-204-C0702 + TSC-202-A0201
  Interventions: Biological: TSC-204-C0702 + TSC-202-A0201
- T-Plex Combination Cohort C+ G (Experimental): TSC-200-A0201 + TSC-202-A0201
  Interventions: Biological: TSC-200-A0201 + TSC-202-A0201
- T-Plex Combination Cohort D + G (Experimental): TSC-203-A0201 + TSC-202-A0201
  Interventions: Biological: TSC-203-A0201 + TSC-202-A0201
- T-Plex Combination Cohort E + G (Experimental): TSC-204-A0101 + TSC-202-A0201
  Interventions: Biological: TSC-204-A0101 + TSC-202-A0201
- T-Plex Combination Cohort F + G (Experimental): TSC-201-B0702 + TSC-202-A0201
  Interventions: Biological: TSC-201-B0702 + TSC-202-A0201

INTERVENTIONS:
Biological: TSC-204-A0201 — Escalating doses of TSC-204-A0201 as a monotherapy
  Arms: Monotherapy Cohort A
Biological: TSC-204-C0702 — Escalating doses of TSC-204-C0702 as a monotherapy
  Arms: Monotherapy Cohort B
Biological: TSC-200-A0201 — Escalating doses of TSC-200-A0201 as a monotherapy
  Arms: Monotherapy Cohort C
Biological: TSC-204-A0201 + TSC-204-C0702 — Escalating doses of TSC-204-A0201 in combination with TSC-204-C0702
  Arms: T-Plex Combination Cohort A + B
Biological: TSC-204-A0201 + TSC-200-A0201 — Escalating doses of TSC-204-A0201 in combination with TSC-200-A0201
  Arms: T-Plex Combination Cohort B + C
Biological: TSC-204-C0702 + TSC-200-A0201 — Escalating doses of TSC-204-C0702 in combination with TSC-200-A0201
  Arms: T-Plex Combination Cohort A + C
Biological: TSC-204-A0201 + TSC-203-A0201 — Escalating doses of TSC-204-A0201 in combination with TSC-203-A0201
  Arms: T-Plex Combination Cohort A + D
Biological: TSC-204-C0702 + TSC-203-A0201 — Escalating doses of TSC-204-C0702 in combination with TSC-203-A0201
  Arms: T-Plex Combination Cohort B + D
Biological: TSC-200-A0201 + TSC-203-A0201 — Escalating doses of TSC-200-A0201 in combination with TSC-203-A0201
  Arms: T-Plex Combination Cohort C + D
Biological: TSC-203-A0201 — Escalating doses of TSC-203-A0201 as a monotherapy
  Arms: Monotherapy Cohort D
Biological: TSC-204-A0101 — Escalating doses of TSC-204-A0101 as a monotherapy
  Arms: Monotherapy Cohort E; T-Plex Combination Cohort E + F
Biological: TSC-201-B0702 — Escalating doses of TSC-201-B0702 as a monotherapy
  Arms: Monotherapy Cohort F; T-Plex Combination Cohort E + F
Biological: TSC-204-A0201 + TSC-204-A0101 — Escalating doses of TSC-204-A0201 in combination with TSC-204-A0101
  Arms: T-Plex Combination Cohort A + E
Biological: TSC-204-A0201 + TSC-201-B0702 — Escalating doses of TSC-204-A0201 in combination with TSC-201-B0702
  Arms: T-Plex Combination Cohort A + F
Biological: TSC-204-C0702 + TSC-204-A0101 — Escalating doses of TSC-204-C0702 in combination with TSC-204-A0101
  Arms: T-Plex Combination Cohort B + E
Biological: TSC-204-C0702 + TSC-201-B0702 — Escalating doses of TSC-204-C0702 in combination with TSC-201-B0702
  Arms: T-Plex Combination Cohort B + F
Biological: TSC-200-A0201 + TSC-204-A0101 — Escalating doses of TSC-200-A0201 in combination with TSC-204-A0101
  Arms: T-Plex Combination Cohort C + E
Biological: TSC-200-A0201 + TSC-201-B0702 — Escalating doses of TSC-200-A0201 in combination with TSC-201-B0702
  Arms: T-Plex Combination Cohort C + F
Biological: TSC-203-A0201 + TSC-204-A0101 — Escalating doses of TSC-203-A0201 in combination with TSC-204-A0101
  Arms: T-Plex Combination Cohort D + E
Biological: TSC-203-A0201 + TSC-201-B0702 — Escalating doses of TSC-203-A0201 in combination with TSC-201-B0702
  Arms: T-Plex Combination Cohort D + F
Biological: TSC-202-A0201 — Escalating doses of TSC-202-A0201 as a monotherapy
  Arms: Monotherapy Cohort G
Biological: TSC-204-A0201 + TSC-202-A0201 — Escalating doses of TSC-204-A0201 in combination with TSC-202-A0201
  Arms: T-Plex Combination Cohort A + G
Biological: TSC-204-C0702 + TSC-202-A0201 — Escalating doses of TSC-204-C0702 in combination with TSC-202-A0201
  Arms: T-Plex Combination Cohort B + G
Biological: TSC-200-A0201 + TSC-202-A0201 — Escalating doses of TSC-200-A0201 in combination with TSC-202-A0201
  Arms: T-Plex Combination Cohort C+ G
Biological: TSC-203-A0201 + TSC-202-A0201 — Escalating doses of TSC-203-A0201 in combination with TSC-202-A0201
  Arms: T-Plex Combination Cohort D + G
Biological: TSC-204-A0101 + TSC-202-A0201 — Escalating doses of TSC-204-A0101 in combination with TSC-202-A0201
  Arms: T-Plex Combination Cohort E + G
Biological: TSC-201-B0702 + TSC-202-A0201 — Escalating doses of TSC-201-B0702 in combination with TSC-202-A0201
  Arms: T-Plex Combination Cohort F + G

SUMMARY:
TScan Therapeutics is developing cellular therapies across multiple solid tumors in which autologous participant-derived engeneered T cells are engineered to express a T cell receptor that recognizes cancer-associated antigens presented on specific Human Leukocyte Antigen (HLA) molecules.

This is a multi-center, non-randomized, multi-arm, open-label, basket study evaluating the safety and preliminary efficacy of single and repeat dose regimens of TCR'Ts as monotherapies and as T-Plex combinations after lymphodepleting chemotherapy in participants with locally advanced, metastatic solid tumors disease.

DETAILED DESCRIPTION:
Participants will be screened in a separate screening study, TSCAN-003 (NCT05812027), to assess their HLA type, tumor-associated antigen (TAA) expression and loss of heterozygosity (LOH) status. The results of these tests will be used to determine initial eligibility in this study.

Depending on the genetic type, participants will be assigned to one of the following study groups:

Monotherapy:

* COHORT A: TSC-204-A0201 targeting MAGE-A1 on HLA-A*02:01
* COHORT B: TSC-204-C0702 targeting MAGE-A1 on HLA-C*07:02
* COHORT C: TSC-200-A0201 targeting HPV16 E7 on HLA-A*02:01
* COHORT D: TSC-203-A0201 targeting PRAME on HLA-A*02:01
* COHORT E: TSC-204-A0101 targeting MAGE-A1 on HLA-A*01:01
* COHORT F: TSC-201-B0702 targeting MAGE-C2 on HLA-B*07:02
* COHORT G: TSC-202-A0201 targeting MAGE-A4 on HLA-A*02:01

T-Plex Combination:

* COHORT AB: TSC-204-A0201 + TSC-204-C0702
* COHORT AC: TSC-204-A0201 + TSC-200-A0201
* COHORT AD: TSC-204-A0201 + TSC-203-A0201
* COHORT AE: TSC-204-A0201 + TSC-204-A0101
* COHORT AF: TSC-204-A0201 + TSC-201-B0702
* COHORT BC: TSC-204-C0702 + TSC-200-A0201
* COHORT BD: TSC-204-C0702 + TSC-203-A0201
* COHORT BE: TSC-204-C0702 + TSC-204-A0101
* COHORT BF: TSC-204-C0702 + TSC-201-B0702
* COHORT CD: TSC-200-A0201 + TSC-203-A0201
* COHORT CE: TSC-200-A0201 + TSC-204-A0101
* COHORT CF: TSC-200-A0201 + TSC-201-B0702
* COHORT DE: TSC-203-A0201 + TSC-204-A0101
* COHORT DF: TSC-203-A0201 + TSC-201-B0702
* COHORT EF: TSC-204-A0101 + TSC-201-B0702
* COHORT AG: TSC-204-A0201 + TSC-202-A0201
* COHORT BG: TSC-204-C0702 + TSC-202-A0201
* COHORT CG: TSC-200-A0201 + TSC-202-A0201
* COHORT DG: TSC-203-A0201 + TSC-202-A0201
* COHORT EG: TSC-204-A0101 + TSC-202-A0201
* COHORT FG: TSC-201-B0702 + TSC-202-A0201

Participants will undergo leukapheresis to collect cells to manufacture the TCR-T products. They will then undergo lymphodepletion and receive one or two doses of the TCR-T cell therapy product as a monotherapy or part of a combination of TCR-Ts (referred to as T-Plex combinations in this study).

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years.
2. Locally advanced (unresectable) or metastatic solid tumor for which there are no available curative treatment options, after failure of the standard of care systemic therapies for that particular indication.
3. Solid tumors, including but not limited to non-nasopharyngeal head and neck cancer, non-small cell lung cancer, cutaneous melanoma, cervical cancer, ovarian cancer, anal cancer and genital cancers. Other tumor types may be permitted if approved by TScan.
4. Participants must express one of the following HLA types, as assessed by a qualified genomics assay in screening study TSCAN-003: HLA-B*07:02, HLA-A*01:01, HLA-C*07:02 and/or HLA-A*02:01
5. Tumor must express one or more of the following: MAGE-A1, MAGE-A4, MAGE-C2, PRAME and HPV16 assessed in the last 8 months in screening study TSCAN-003 (NCT05812027).
6. Eastern Cooperative Oncology Group (ECOG) Performance status 0-1 at screening.
7. Participants must be able to understand and be willing to give informed consent; decision-impaired adults may consent with their legally authorized representative.
8. At least 1 measurable lesion per modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
9. Adequate bone marrow and organ function.

Exclusion Criteria:

1. Medical or psychological conditions that would make the participant unsuitable candidate for cell therapy at the discretion of the PI.
2. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, cardiac arrhythmia requiring antiarrhythmic or procedure, or other clinically significant cardiac disease within 12 months of enrollment
3. Have a history of ASTCT Grade 4 CRS, Grade 3 or greater ICANS, or Grade 3 or greater IECHS. Participants with a history of lower grade CRS, ICANS, or IECHS may be eligible, pending review and approval by the Medical Monitor.
4. History of stroke or transient ischemic attack (TIA) within 6 months of enrollment
5. Systemic corticosteroid therapy >10 mg of prednisone daily or equivalent within 7 days of enrollment.
6. History of severe hypersensitivity to fludarabine or cyclophosphamide or study product excipients including human serum albumin, Cryostor (DMSO or Dextran 40), or Plasma-Lyte.
7. Untreated or symptomatic central nervous system (CNS) metastases or cytology proven carcinomatous meningitis.
8. Concurrent receipt of another anti-cancer therapy. Have a history of acute mental status changes of unknown etiology within 6 months prior to enrollment, or any neurological or neurodegenerative disorder (e.g., Parkinson disease, Huntington disease, uncontrolled seizure disorder) that may increase the risk for or confound the assessment of neurotoxicity.
9. Presence of fungal, bacterial, viral, or other infection requiring anti-microbials for management.
10. Tumors that have HLA LOH using a central lab clinical trial assay of HLAs addressed by the monotherapy and/or T-Plex combination TCR-Ts in the protocol and have no available TCR-T options for intact HLAs in the participant's tumor.
11. Participants who regularly require supplemental oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of monotherapy and T- Plex combination TCR-Ts | 28 days
  Number of subjects with dose limiting toxicities (DLT)
Determine the recommended phase 2 dose of monotherapy and T- Plex combination TCR-Ts | Up to 12 months
  Frequency and severity of DLTs, AEs and SAEs

SECONDARY OUTCOMES:
Investigate preliminary anti-tumor activity of monotherapy and T- Plex combination TCR-Ts | Up to 12 months
  Response Evaluation Criteria In Solid Tumors RECIST 1.1
Investigate the feasibility of repeat dosing of monotherapy and T- Plex combination TCR-Ts | Up to 12 months
  Frequency and severity of DLTs, AEs and SAEs

OTHER OUTCOMES:
To measure the persistence of T-Plex TCR-T cells in the peripheral blood with single and repeat doses | Up to 24 months
  Percentage of TCR-T cells in the peripheral blood after single and repeat doses
To measure the infiltration of T-Plex TCR-T cells into tumors in post-treatment biopsies | Up to 24 months
  Percentage of TCR-T cells in the tumor after single and repeat doses
To measure the immune activation markers in the tumor after single and repeated doses | Up to 24 months
  Status of immune activation markers in the tumor after single and repeat doses

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Pinchasik, MD, Study Director — TScan Therapeutics
Locations (21):
- United States (21):
  - HonorHealth Research and Innovation Institute, Scottsdale, Arizona
  - University of California San Diego, San Diego, California
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Healthcare System, Hollywood, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Health, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Allegheny Hospitals Network, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No